CLINICAL TRIAL: NCT02698254
Title: Pilot Trial of Dose-Volume Constraints for Reirradiation of Recurrent Brain Tumors
Brief Title: Radiation Therapy in Treating Patients With Recurrent Brain Tumors Who Have Undergone Previous Radiation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0586; NCI-2016-00536 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0586 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (conventional fractionation) (Experimental): Patients undergo radiation therapy with conventional fractionation and dose constraints. Treatment continues for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Quality-of-Life Assessment; Radiation: Radiation Therapy
- Arm II (conventional fractionation, bevacizumab) (Active Comparator): Patients undergo radiation therapy with conventional fractionation and dose constraints. Patients also receive bevacizumab concurrently at the discretion of the treating neuro-oncologist. Treatment continues for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Bevacizumab
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar SCT501; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
  Arms: Arm II (conventional fractionation, bevacizumab)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy with conventional fractionation
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This pilot clinical trial studies the side effects and best dose of radiation therapy in patients with brain tumors that have come back after previous treatment with radiation therapy. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving radiation therapy in different ways may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the rate of grade 3 or higher central nervous system (CNS) necrosis 6 months after reirradiation of the brain for recurrent tumor.

SECONDARY OBJECTIVES:

I. To evaluate acute and late toxicities of reirradiation. II. To evaluate longitudinal changes in symptom burden of patients undergoing reirradiation.

III. To use Advanced Brain Tumor Imaging (ABTI) to evaluate changes in the brain after reirradiation, including progression, pseudoprogression, and radionecrosis.

IV. To estimate progression-free survival (PFS) and overall survival (OS) following reirradiation.

OUTLINE: Patients are assigned to 1 of 2 arms based on age.

ARM I (Age 0-18 years): Patients undergo radiation therapy with conventional fractionation and dose constraints. Treatment continues for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM II (Age > 18 years): Patients undergo radiation therapy with conventional fractionation and dose constraints. Patients also receive bevacizumab concurrently at the discretion of the treating neuro-oncologist. Treatment continues for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month, then every 2 months for 1 year, then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Previous pathologic confirmation of a tumor treated with radiation to the brain completed at least 6 months prior to the start of planned reirradiation, except for patients with tumors that are routinely diagnosed without biopsy, including germinoma and optic pathway glioma; patients with a history of cranial irradiation for leukemia are eligible
* Patient must have received one and only one previous course of radiation to the brain, delivered at 1.5 - 2.5 Gy/fraction, one fraction per day
* Multidisciplinary evaluation of the patient must be performed with a consensus recommendation for reirradiation
* Patient may not receive concurrent chemotherapy with reirradiation, other than temozolomide or bevacizumab given at the discretion of the treating neuro-oncologist
* Patient must have imaging findings within the last 3 months consistent with recurrent disease in the brain; pathologic diagnosis of recurrence is not required
* Patient may undergo surgical resection prior to reirradiation
* Dose-volume histogram data and cross-sectional imaging from previous radiation must be obtained; electronic dosimetry records in Digital Imaging and Communications in Medicine (DICOM) format from previous radiation are strongly preferred
* Signed informed consent by patient and/or parents or legal guardian
* Lansky/Karnofsky performance status score of 50-100

Exclusion Criteria:

* Patients with recurrent diffuse intrinsic pontine glioma (DIPG)
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Highest grade of central nervous system (CNS) necrosis | At 6 months
  The outcome will be categorized as (death within 6 months), (alive at month 6 with necrosis), (alive at month 6 without necrosis). The probabilities of these outcomes will be estimated using 95% posterior credible intervals assuming a Dirichlet (.33, .33, .33) prior.

SECONDARY OUTCOMES:
Incidence of acute and late toxicities | Up to 3.5 years
Overall survival (OS) time | Up to 3.5 years
  Will be estimated by Kaplan-Meier method, and the relationship of OS to baseline covariates will be evaluated by Bayesian survival time regression.
Progression-free survival (PFS) time | Up to 3.5 years
  Will be estimated by Kaplan-Meier method, and the relationship of PFS to baseline covariates will be evaluated by Bayesian survival time regression.
Quality of life | Up to 3.5 years
  Will be assessed using the MD Anderson Symptom Inventory-Brain Tumor (MDASI-BT) and patient-reported outcomes measurement information system (PROMIS) instrument.
Imaging changes as measured by Advanced Brain Tumor Imaging (ABTI) | Up to 3.5 years

OTHER OUTCOMES:
Symptom burden | Up to 3.5 years
  Will be measured by MDASI-BT questionnaire in adults and PROMIS short forms in children.

CONTACTS AND LOCATIONS:
Overall Officials: Susan L McGovern, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org